CLINICAL TRIAL: NCT01246661
Title: MilkScreen™ Home Test for Alcohol in Breast Milk Clinical Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: UpSpring Baby, Ltd. (Industry)
Responsible Party: Matt Pope, UpSpring Baby
Other Study IDs: 4001-002
Record Dates: First submitted 2010-11-22; First posted 2010-11-23 (Estimated); Last update posted 2010-11-23 (Estimated); Status verified 2010-11

CONDITIONS: Alcohol in Breastmilk

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to evaluate if the UpSpring Milkscreen Alcohol Test works to detect alcohol in breast milk that will be donated during this study. This research is being done because the sponsoring company, UpSpring, wants to determine if this test will work and, if it does, how well it will work to detect levels of alcohol in breast milk.

DETAILED DESCRIPTION:
MilkScreen™ Home Test for Alcohol in Breast Milk is intended as an OTC test for the presence of alcohol in breast milk. This study will obtain data to demonstrate the agreement of MilkScreen™ compared to the reference method, head space Gas Chromatography-Mass Spectrometry (GC-MS) for alcohol content and will additionally provide validation of the usability of the device by the intended users.

The study will use a minimum of 50 lactating mothers who will come into a center in small groups in a contrived social setting like a wine tasting. Upon completion of informed consent and demonstration of meeting inclusion/exclusion criteria, subjects will be tested with disposable breathalyzer test and baseline breast milk samples provided. The baseline breast milk samples will be tested with the test article by the subject. Aliquots from the same samples will be prepared for testing by an outside lab with GC-MS.

Subjects will be asked to provide baseline demographics such as height and weight, days since birth of child, race/ethnicity, and information about any prescription or OTC drugs, herbal compounds or vitamins they have taken in the previous 72 hours.

Subjects will be provided with up to 3 alcoholic beverages over the course of a three to four hour period. At prescribed time intervals following consumption, subjects will be asked to provide a breast milk sample and to submit to a breathalyzer test. Each breast milk sample will be tested by the subject with the test article following the labeling instructions only and the sample will also be aliquoted into tightly sealing, low head space sample containers for method comparison testing by an outside lab with GC-MS.

Subjects will be asked to drink at least one drink, but may ingest up to two additional alcoholic beverages during the course of the study. Each subject's blood alcohol content (BAC) will be monitored before each additional drink is provided and will not be allowed to consume additional drinks if their BAC as measured by the disposable breathalyzer device exceeds 0.10% (100 mg/dL). All drinks will be prepared such that they contain alcohol consistent with a standard alcoholic drink, as defined by the National Institute on Alcohol Abuse and Alcoholism (12 ounces of beer, 8-9 ounces of malt liquor, 5 ounces of table wine, or 1.5 ounces of liquor). Subjects will be asked to self report whether they finished their drink at the point when samples are taken. Subjects will be provided with transportation to and from the study site using designated non-drinking drivers.

Samples of breast milk taken both prior to and following the ingestion of alcohol will be coded and thereby blinded to the lab. The lab will run GC-MS on each specimen and will report the results to the Sponsor. This data will be compared with the data reported by each subject and analyzed to demonstrate that the MilkScreen™ Home Test for Alcohol in Breast Milk agrees to a high degree to the reference method, GC-MS, to support the test article's intended use.

Subjects will be asked to complete a questionnaire on the usability of the labeling instructions on MilkScreen™ Home Test for Alcohol in Breast Milk to demonstrate that consumers can use the directions properly to test their breast milk for the presence of alcohol and properly interpret the results.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age equal to or greater than 21 years
* Actively breast-feeding
* Willing to drink at least one alcoholic beverage (wine or beer) during study in a controlled setting
* Willing to arrive to the study session prior to consuming any alcoholic beverages within the last 24 hours.
* Willing to attend single session study for 3-4 hours duration until their BAC drops below 0.06%
* Willing to accept designated driver or study-supplied transportation
* Willing to agree to not breast feed their infant for 2 hours following departure from the study session
* English language fluency

Exclusion Criteria:

* Distance of more than 25 miles from study site
* Pregnant (pregnancy test will be administered at time of study)
* Communicable diseases (e.g., Flu)
* HIV Positive
* History of Alcoholism
* Arriving to the study session with a BAC at or above 0.01%
* Any medical condition which precludes the subject from drinking alcohol
* Skilled or trained in clinical laboratory procedures

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female subjects 21 years and older will be recruited for this study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-04 (Actual); Study Completion 2010-11 (Estimated)